CLINICAL TRIAL: NCT03369834
Title: Acute Effect of Light-emitting Diode-phototherapy on Strength, Functional Performance and Blood Flow in Diabetic Subjects
Brief Title: Light-emitting-diode in Diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rinaldo Roberto de Jesus Guirro (Other)
Responsible Party: Sponsor-Investigator, Rinaldo Roberto de Jesus Guirro, Clinical Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1143-3534
Record Dates: First submitted 2017-11-30; First posted 2017-12-12 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Neuropathies
Keywords: phototherapy; diabetes mellitus; exercise
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Intervention Model Description: Control Group (GC=13) LED red group (GLED-V = 13) Infrared LED Group (GLED-IV = 13) Mixed Group (GM = 13) Sham Group (GP = 13)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control Group (No Intervention): the volunteers of this group will not be submitted to the intervention.
- Red LED group (Experimental): in the volunteers of this group will be applied Red Light-emitting diode device with the length 620nm wave along the entire tibialis anterior muscle and bilateral sural triceps.
  Interventions: Device: Red Light-emitting diode device
- LED group infrared (Active Comparator): in the volunteers of this group will be applied Infrared Light-emitting diode device with the wavelength of 940nm throughout the tibialis anterior muscle and bilateral sural triceps.
  Interventions: Device: Infrared Light-emitting diode device
- LED group mixed (Active Comparator): in the volunteers of this group will be applied Infrared and Red Light-emitting diode device with the wavelength of 940nm and 620nm throughout the tibialis anterior muscle and bilateral sural triceps.
  Interventions: Device: Infrared and Red Light-emitting diode device
- Sham Group (Placebo Comparator): LED device off.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Red Light-emitting diode device — The phototherapy will be applied for 3 days followed by a red LED blanket of 25x40 cm2, with equidistant distribution - 1 cm between them, with total energy per area of 180 J, bilaterally on the anterior tibial and triceps sural muscles, bilaterally. The intervention of these muscular groups is made possible by the distal involvement of diabetic polyneuropathy.
  All LEDs will be checked at the beginning of the project in the Laboratory of Photophysics of the Faculty of Philosophy, Sciences and Letters of Ribeirão Preto, University of São Paulo, in which the wavelengths will be checked, the angle of radiation, power and power density.
  Arms: Red LED group
Device: Infrared Light-emitting diode device — The phototherapy will be applied for 3 days followed by a infrared LED blanket of 25x40 cm2, with equidistant distribution - 1 cm between them, with total energy per area of 180 J, bilaterally on the anterior tibial and triceps sural muscles, bilaterally. The intervention of these muscular groups is made possible by the distal involvement of diabetic polyneuropathy.
  All LEDs will be checked at the beginning of the project in the Laboratory of Photophysics of the Faculty of Philosophy, Sciences and Letters of Ribeirão Preto, University of São Paulo, in which the wavelengths will be checked, the angle of radiation, power and power density.
  Arms: LED group infrared
Device: Infrared and Red Light-emitting diode device — The phototherapy will be applied for 3 days followed by a infrared and Red LED blanket of 25x40 cm2, with equidistant distribution - 1 cm between them, with total energy per area of 180 J, bilaterally on the anterior tibial and triceps sural muscles, bilaterally. The intervention of these muscular groups is made possible by the distal involvement of diabetic polyneuropathy.
  All LEDs will be checked at the beginning of the project in the Laboratory of Photophysics of the Faculty of Philosophy, Sciences and Letters of Ribeirão Preto, University of São Paulo, in which the wavelengths will be checked, the angle of radiation, power and power density.
  Arms: LED group mixed
Device: Sham — LED device off.
  Arms: Sham Group

SUMMARY:
Diabetes mellitus (DM) is a metabolic disorder, characterized by hyperglycemia and metabolic disorders, resulting in changes in insulin secretion and / or action. Physical function is critical for functional independence, and chronic diseases such as diabetes can lead to functional decline, and diabetes mellitus is a major contributor to the progression of sarcopenia and physical disability. DM is also known to have a strong associated with the development of peripheral arterial disease. Peripheral arterial disease is characterized by obstruction of the arteries of the lower limbs, leading to a low oxygenation of the muscles of the lower extremities. Among the physiotherapeutic resources that can be used, phototherapy involves the use of light for the treatment of muscular injuries, by modulating the physiological processes associated with the repair process. Clinical trials show that light emitting diode (LED) is a technique that interferes with muscle strength, generating an increase in maximal voluntary contraction and peak torque. It is hypothesized that the LED application is capable of improving the muscular strength, fatigue, functional performance and blood flow capabilities in individuals with diabetes. It is also expected that the results of this study may contribute to and increase the resources used by physiotherapists within the clinical scope, contributing to the care of diabetic patients.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a metabolic disorder, characterized by hyperglycemia and metabolic disorders, resulting in changes in insulin secretion and / or action. Physical function is critical for functional independence, and chronic diseases such as diabetes can lead to functional decline, and diabetes mellitus is a major contributor to the progression of sarcopenia and physical disability. DM is also known to have a strong associated with the development of peripheral arterial disease. Peripheral arterial disease is characterized by obstruction of the arteries of the lower limbs, leading to a low oxygenation of the muscles of the lower extremities. Among the physiotherapeutic resources that can be used, phototherapy involves the use of light for the treatment of muscular injuries, by modulating the physiological processes associated with the repair process. Clinical trials show that LED is a technique that interferes with muscle strength, generating an increase in maximal voluntary contraction and peak torque. It is hypothesized that the LED application is capable of improving the muscular strength, fatigue, functional performance and blood flow capabilities in individuals with diabetes. It is also expected that the results of this study may contribute to and increase the resources used by physiotherapists within the clinical scope, contributing to the care of diabetic patients. A randomized and blinded clinical trial will be carried out at the Physiotherapeutic Resources Laboratory (LARF) of the University of São Paulo Medical School of Ribeirão Preto (FMRP-USP). The study procedures will be performed in 5 days. On the first day (pre-treatment), the volunteers will be evaluated for functionality (Time Up and Go), cardiopulmonary capacity (6-minute walk test), evaluation of muscle function (isokinetic dynamometer), neuromuscular recruitment (electromyography) gastrocnemius and evaluation of blood flow (Doppler) of the tibial and popliteal arteries. On the second, third and fourth day volunteers of GLED-V, GLED-IV, GM e GP will return to the application of LED intervention according to the group in which they are allocated. On the fifth day (reevaluation) the volunteers will perform the same tests of the first day.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary and insufficiently active individuals with the the International Physical Activity Questionnaire (IPAQ) .
* Both sexes
* Age range of 45 to 70 years
* Diagnostic Scale for Diabetic Distal Polyneuropathy - Score 3 or more

Exclusion Criteria:

* Present musculoskeletal or neurological lesions that make it impossible to perform the functional and strength tests.
* Negative result for the tactile sensitivity test with the monofilament.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
strength capacities | Twenty minutes
  N/m

SECONDARY OUTCOMES:
Electromyography | Twenty minutes
  Muscle recruitment - Hertz
Time up and Go | two minutes
  time
6-minute walk test | ten minutes
  meters
blood flow | ten minutes
  mL/s

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo RJ Guirro, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Toma RL, Vassao PG, Assis L, Antunes HK, Renno AC. Low level laser therapy associated with a strength training program on muscle performance in elderly women: a randomized double blind control study. Lasers Med Sci. 2016 Aug;31(6):1219-29. doi: 10.1007/s10103-016-1967-y. Epub 2016 Jun 1. PMID 27250715
- See also: access platform — https://www.ncbi.nlm.nih.gov/pubmed/?term=Low+level+laser+therapy+associated+with+a+strength+training+program+on+muscle+performance+in+elderly+women%3A+a+randomized+double+blind+control+study.